CLINICAL TRIAL: NCT03202680
Title: A Randomized, Controlled-Feeding, Crossover Trial to Assess the Effects of Increasing Lean Beef Consumption Within a Healthy Dietary Pattern on Insulin Sensitivity in Men and Women With Risk Factors for Diabetes Mellitus.
Brief Title: Lean Beef Consumption and Insulin Sensitivity in Men and Women With Risk Factors for Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: MB-1606
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Metabolic Syndrome; PreDiabetes
MeSH Terms: conditions — Metabolic Syndrome; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- USDA Style Diet (Active Comparator): Healthy, low saturated fat, United States Department of Agriculture (USDA) style diet.
  Interventions: Other: USDA Style Diet
- Lean Beef Diet (Experimental): Healthy, low saturated fat, high in lean beef diet.
  Interventions: Other: Lean Beef Diet

INTERVENTIONS:
Other: USDA Style Diet — USDA style healthy diet, low in saturated fats.
  Arms: USDA Style Diet
Other: Lean Beef Diet — A lean beef containing healthy diet, low in saturated fats.
  Arms: Lean Beef Diet

SUMMARY:
The objective of this trial is to compare the effects of a healthy, lean beef diet and an average American, United States Department of Agriculture (USDA) style diet, that is low in saturated fatty acids (SFA), on insulin sensitivity in men and women with risk factors for diabetes mellitus.

DETAILED DESCRIPTION:
This is a randomized, controlled, crossover study that includes two screening visits, one baseline visit, two 28-d test periods and an end-of-washout visit. A 2-week washout period will separate the two treatments. Subjects will be screened to identify metabolic syndrome and/or prediabetes at the screening visits. Eligible subjects will be randomly assigned to a test sequence (USDA/lean beef or lean beef/USDA diets) and the appropriate calorie menu within each test diet, which will be determined based on each subject's calculated energy needs for weight maintenance. Study foods will be dispensed, and subjects will be instructed to consume all of the foods in their entirety for the duration of each 28-d test period, and avoid consuming any additional food or drink items that has not been provided to them. Compliance will be assessed through a Food Deviation Log where subjects will record any non-study food/beverages consumed, and any portions of the study foods not consumed.

An intravenous glucose tolerance test (IVGTT) will be completed at baseline and the end of each treatment period, and fasting glucose and insulin will also be measured at screening and at the first test visit in each treatment period. Fasting blood samples will be collected for lipid profile and high-sensitivity C-reactive protein (hs-CRP) measurements at all treatment visits. Additionally, fasting blood will be drawn for measurement of apolipoprotein B and A1 and lipoprotein particles and subfractions at baseline and the end of each treatment period.

Assessments of vital signs, body weight, evaluation of inclusion and exclusion criteria, medication/supplement use, and adverse effects will be performed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. BMI of 25.0-39.9 kg/m2.
2. Metabolic syndrome (exhibiting at least 3 out of 5 of the criteria) AND/OR prediabetes (either fingerstick glycated hemoglobin 5.7-6.4%, fasting fingerstick capillary glucose of 100-125 mg/dL, or 2-h post-prandial glucose of 140-199 mg/dL).
3. Fasting LDL-C level <200 mg/dL and fasting TG level <400 mg/dL.
4. Willingness to consume only study-related foods/beverages during each test period and consume all of the study foods provided for each day.
5. Willingness to come to the clinic for study food pick-up as needed.
6. Judged to be in general good health, aside from the inclusionary metabolic criteria for the study, on the basis of medical history and screening laboratory tests.

Exclusion Criteria:

1. Atherosclerotic cardiovascular disease including any of the following: clinical signs of atherosclerosis including peripheral arterial disease, abdominal aortic aneurysm, carotid artery disease [symptomatic (e.g., transient ischemic attack or stroke of carotid origin) or >50% stenosis on angiography or ultrasound], history of myocardial infarction, angina, or other forms of clinical atherosclerotic disease (e.g., renal artery disease).
2. History or presence of clinically important pulmonary (including uncontrolled asthma), endocrine (including type 1 or type 2 diabetes mellitus), chronic inflammatory disease (including irritable bowel disease, lupus, rheumatoid arthritis), hepatic, renal, hematologic, immunologic, dermatologic, neurologic, psychiatric, or biliary disorders.
3. Known allergy, sensitivity, or intolerance to any ingredients in the study foods (e.g., dairy, nuts, etc.).
4. Uncontrolled hypertension.
5. Recent history of cancer except for non-melanoma skin cancer.
6. Recent change in body weight of ± 4.5 kg (10 lbs).
7. Unstable use of any antihypertensive medication.
8. Recent use of medications intended to alter the lipid profile [e.g., bile acid sequestrants, cholesterol absorption inhibitor, fibrates, niacin (drug form), omega-3-ethyl ester drugs, and/or proprotein convertase subtilisin kexin type 9 (PCSK9) inhibitors], weight-loss drugs or programs, systemic corticosteroid drugs, medications known to influence carbohydrate metabolism (e.g., adrenergic receptor blockers, diuretics, and/or hypoglycemic medications).
9. Recent use of foods or dietary supplements known to influence lipid metabolism (e.g., omega-3 fatty acids supplements or fortified foods, sterol/stanol products, red rice yeast supplements, garlic supplements, soy isoflavone supplements, niacin or its analogues at doses >400 mg/d and irregular or inconsistent use of Metamucil® or viscous fiber-containing supplements.
10. Recent use of antibiotics.
11. Pregnant, planning to be pregnant during the study period, lactating, or of childbearing potential and unwilling to commit to the use of a medically approved form of contraception throughout the study period.
12. Extreme dietary habits (e.g., very low carbohydrate diet, vegan, vegetarian, etc.) or unwillingness to consume study foods.
13. Current or recent history or strong potential for drug or alcohol abuse.
14. History of a diagnosed eating disorder (e.g., anorexia or bulimia nervosa).
15. Recent exposure to any non-registered drug product.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity index (Si) | Up to 50 minutes - measured at baseline, and end of each treatment period.
  Differences in the change from baseline between test conditions (lean beef diet and USDA diet) in the insulin sensitivity index (Si) using the short IVGTT.

SECONDARY OUTCOMES:
Disposition index of pancreatic beta-cell function [Si x acute insulin response to intravenous glucose (AIRg)] | Up to 50 minutes - measured at baseline, and end of each treatment period.
  Percent change (or change) from baseline to the end of each test condition.
Fractional glucose disappearance constant from t = 10-50 min (Kg) | Up to 50 minutes - measured at baseline, and end of each treatment period.
  Percent change (or change) from baseline to the end of each test condition.
Homeostasis model assessment of beta cell function (HOMA%B) and insulin sensitivity (HOMA%S) | Up to 28 days for each treatment period.
  Percent change (or change) from baseline to the end of each test condition.
Insulin sensitivity (HOMA%S) | Up to 28 days for each treatment period.
  Percent change (or change) from baseline to the end of each test condition.
Total Cholesterol (TC) | Up to 28 days for each treatment period.
  Percent change (or change) in TC from baseline to the end of each test condition
Low-density Lipoprotein Cholesterol (LDL-C) | Up to 28 days for each treatment period.
  Percent change (or change) in LDL-C from baseline to the end of each test condition
High-density Lipoprotein Cholesterol (HDL-C) | Up to 28 days for each treatment period.
  Percent change (or change) in HDL-C from baseline to the end of each test condition
Non-HDL-C | Up to 28 days for each treatment period.
  Percent change (or change) in Non-HDL-C from baseline to the end of each test condition
Triglycerides (TG) | Up to 28 days for each treatment period.
  Percent change (or change) in TG from baseline to the end of each test condition
TC/HDL-C ratio | Up to 28 days for each treatment period.
  Percent change (or change) in TC/HDL-C ratio from baseline to the end of each test condition
High-sensitivity C-reactive protein (hs-CRP) | Up to 28 days for each treatment period.
  Percent change (or change) from baseline to the end of each test condition in levels of hs-CRP
Resting, seated systolic and diastolic blood pressures | Up to 28 days for each treatment period.
  Percent change (or change) from baseline to the end of each test condition.
Lipoprotein subfraction and particle concentrations. | Up to 28 days for each treatment period.
  Percent change (or change) in lipoprotein subfraction and particle concentrations from baseline to the end of each test condition.
Apo B measurements. | Up to 28 days for each treatment period.
  Percent change (or change) in Apo B levels from baseline to the end of each test condition.
Apo A1 measurements. | Up to 28 days for each treatment period.
  Percent change (or change) in Apo A1 levels from baseline to the end of each test condition.

CONTACTS AND LOCATIONS:
Locations (1):
- MB Clinical Research, LLC, Boca Raton, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maki KC, Wilcox ML, Dicklin MR, Buggia M, Palacios OM, Maki CE, Kramer M. Substituting Lean Beef for Carbohydrate in a Healthy Dietary Pattern Does Not Adversely Affect the Cardiometabolic Risk Factor Profile in Men and Women at Risk for Type 2 Diabetes. J Nutr. 2020 Jul 1;150(7):1824-1833. doi: 10.1093/jn/nxaa116. PMID 32359153